CLINICAL TRIAL: NCT05829707
Title: Long-term Outcomes of Breast Cancer Patients Receiving Levobupivacaine Wound Infiltration or Diclofenac for Postoperative Pain Relief
Brief Title: Long-term Outcomes of Breast Cancer Patients After Wound Infiltration Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Osijek University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OsijekUH21
Record Dates: First submitted 2023-04-12; First posted 2023-04-26 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Analgesia; Hand Strength; Health Related Quality of Life; Chronic Shoulder Pain; Breast Cancer Female; Surgical Wound Infiltration; Lymph Node Dissection
Keywords: Acute Postoperative Pain; Breast Cancer; Postoperative analgesia; Patient-Controlled Analgesia; Levobupivacaine; Diclofenac; Hand Grip Strength; Quality of life; Treatment Outcome
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms | interventions — Diclofenac; Anti-Inflammatory Agents, Non-Steroidal; Anesthetics, Local

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: On the one-year control examination, the investigator was blinded on the type of postoperative analgesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Diclofenac (Active Comparator): All patients underwent quadrantectomy or mastectomy with axillary lymph node dissection. They received diclofenac 2 x 75 mg intravenously on the first day after surgery. During the 3 subsequent days, from day 2 to day 4 postoperatively patients were given 3 x 50 mg diclofenac tablets orally. The medicine was delivered by the nurse, and the patients drank tablets in front of her.
  Interventions: Drug: Diclofenac Sodium
- Levobupivacaine bolus analgesia (Experimental): Group Levobupivacaine Bolus received 0.5 mg/kg 0.5% Levobupivacaine HCl every 8 h via wound catheter. The dose of levobupivacaine was prescribed by the doctor and the drug was delivered by the nurse.
  Interventions: Drug: Levobupivacaine bolus analgesia
- Levobupivacaine PCA group (Experimental): Group Levobupivacaine patient-controlled analgesia (PCA) received 0.05 mg/kg 0.5% Levobupivacaine HCl continuously via wound catheter delivered by CADD - Legacy® PCA Pump. These patients were allowed to add a dose of 7.5 mg 0.5% levobupivacaine in case of pain by pressing the patient's button on the PCA pump, with a lock-out period of 4 hours.
  Interventions: Drug: Levobupivacaine PCA group

INTERVENTIONS:
Drug: Diclofenac Sodium — A group of patients with breast cancer who were randomized to the diclofenac group by drawing random numbers was given 2 x 75 mg of drug IV on the first PO day and then 3 x 50 mg tablets orally for postoperative analgesia.
  All patients were assessed before the surgical procedure: hand grip strength, shoulder disability, and health-related quality of life were measured. Pain relief was assessed by the visual analog scale (VAS) from 0-10.
  Rescue analgesia was offered for pain >4 on the VAS, meperidine 20-30 mg for VAS >or = 4
  Other Names: Nonsteroidal antiinflammatory drug
  Arms: Diclofenac
Drug: Levobupivacaine bolus analgesia — The levobupivacaine dose was calculated by a doctor. A wound infiltration catheter was inserted at the end of the surgical procedure by a surgeon. A first dose of local anesthetic was delivered at the end of the surgical procedure to test catheter placement. Bolus doses of local anesthetics based on the patients' body weight were thereafter delivered by the nurse in 8 hours intervals.
  All patients were assessed before the surgical procedure and hand grip strength, shoulder disability, and health-related quality of life were measured. Pain relief was assessed by the visual analog scale (VAS) from 0-10.
  Rescue analgesia was offered for pain >4 on the VAS, meperidine 20-30 mg for VAS >or = 4.
  Other Names: Postoperative wound infiltration with bolus applications of local anesthetic, Chirocaine 0.5%
  Arms: Levobupivacaine bolus analgesia
Drug: Levobupivacaine PCA group — The levobupivacaine dose was calculated by a doctor. A wound infiltration catheter was inserted at the end of the surgical procedure by a surgeon. Levobupivacaine was delivered by PCA pump (CADD - Legacy® PCA Pump, Model 6300, Smiths Medical MD, Inc., St. Paul, USA). A drug delivery was started at the end of the surgical procedure.
  All patients were assessed before the surgical procedure: hand grip strength, shoulder disability, and health-related quality of life were measured. Pain relief was assessed by the visual analog scale (VAS) from 0-10.
  Rescue analgesia was offered for persisting pain >4 on the VAS, and meperidine 20-30 mg for VAS >or = 4.
  Other Names: Postoperative continuous wound infiltration analgesia with local anesthetic, Chirocaine 0.5%
  Arms: Levobupivacaine PCA group

SUMMARY:
In the study that was conducted from 05.01.2009 - 31.12.2012. 120 patients were examined. By drawing random numbers, the patients were randomized into 3 groups for postoperative analgesia:

1. Diclofenac 2 mg/kg/day - control,
2. Wound infiltration via wound catheter with catheter tip placed in the axilla, 3*0.5 mg/kg 0.5% levobupivacaine bolus dose.
3. 0.05 mg/kg/h 0.5% levobupivacaine continuously via wound infiltration catheter with catheter tip placed in the axilla. The drug was delivered using a PCA pump for 24 hours.

The aim was to compare early postoperative outcomes - pain control on a visual analog scale of 1-10, hand grip strength, and quality of life after surgery and after 1 year.

Long-term survival was examined subsequently, from the hospital register.

DETAILED DESCRIPTION:
Before the operation, the patients were randomized into 3 groups: the first group received diclofenac for postoperative analgesia. On the first day, they received 2 x 75 mg intravenously, and then 3 x 50 mg tablets. For the wound infiltration with levobupivacaine, a perforated catheter was placed at the end of the surgical procedure by the surgeon in both groups of patients. The tip of the catheter was in the axillary fossa, where the dissection was performed. Patients in the levobupivacaine bolus group (N=39) received three times a day bolus doses of 0.5 mg/kg 0.5% levobupivacaine (Chirocaine, Abbot S.p.A., Latina, Italy) through the catheter. The dose of levobupivacaine was prescribed by the doctor, and the drug was delivered by the nurse. In levobupivacaine, PCA group (N=40) women had the same catheter placed, but received 0.05 mg/kg/h 0.5% levobupivacaine continuously for 24 hours via a catheter placed in the axilla. Levobupivacaine was delivered by PCA pump (CADD - Legacy® PCA Pump, Model 6300, Smiths Medical MD, Inc., St. Paul, USA). These patients were allowed to add a dose of 7.5 mg 0.5% levobupivacaine in case of pain by pressing the patient's button on the PCA pump, with a lock-out period of 4 hours. Postoperative pain was measured with a visual analog scale (VAS). All patients had the option of additional analgesia, using NSAIDs for pain <4 or meperidine for VAS >4. After the surgery, the patients received oncological chemoradiotherapy, depending on the type and stage of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients whose disease requires axillary lymph node dissection
* who consented to participate in the study
* aged 30 - 75
* The patient is able to understand all three methods of analgesia
* Patients can receive any of the study drugs
* Able to understand and complete questionnaires on quality of life and shoulder pain

Exclusion Criteria:

* Age <30 years - >75 years
* Patients who refused to participate in the study (at any stage of the study)
* Patients who after histological analysis did not require axillary lymph node dissection
* Patients with known intolerance to study drugs
* Patients who unintentionally removed wound infiltration catheters.
* Patients who required surgical reintervention during the study period
* Patients having adverse reactions to any study drug.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patients were included in the study
Enrollment: 120 (Actual)
Dates: Start 2009-01-05 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | from 1-4 days postoperative, day of surgery is day 1
  Pain after mastectomy was evaluated by self-reports from patients using a Visual Analog Scale (VAS) from 0 - no pain up to 10 - the worst pain imaginable.
Hand grip strength | Before surgery, on day 4 after surgery, and one year after surgery
  Hand grip strength (HGS) was measured preoperatively, 4 days after surgery and at follow-up after 1 year, using a handheld dynamometer (Dynatest®, Rud. Reister Gmbh&CaKG, Jungingen, Germany) and expressed in bars. Mean expected normal values for female patients are in the range between 0.4-0.6 bar.
Shoulder disability | Before surgery and after one year at surgical control.
  Shoulder pain was assessed using the Shoulder Disability Questionnaire (SDQ), and shoulder pain was assessed in 16 typical situations such as writing, opening a door, sleeping on the operated side, or carrying a load. The maximal score was all positive ( 16 in 16, 100%), suggesting that pain was present in all 16 clinical situations, and the minimum score is 0 (0 positive responses /16 situations, 0% - no disability in any situation.
Health related quality of life | Before surgery and after one year at surgical control.
  Health-related quality of life was assessed using the Croatian version of the SF-36 questionnaire. There were eight domains examined: physical health, role limitation due to physical problems, pain, general health perception, energy / vitality, social functioning, limitations due to emotional problems, and general mental health.
  This instrument summarizes health perception from the patient's perspective. SF-36 scores range from 0 (worst) to 100 (best) (5).

SECONDARY OUTCOMES:
Long-term survival - 5 years after surgery | Five years after surgery
  Survival after 5 years from the surgery will be checked through the hospital registry, or for those who died through the official population records and death registers of the Republic of Croatia. Patients' outcomes are dichotomous and are presented as alive or dead 5 years after surgery.
Long term survival - 10 years after surgery | Ten years after surgery until data were collected
  Survival after 10 years from the surgery will be checked through the hospital registry, or for those who died through the official population records and death registers of the Republic of Croatia. Patients' outcomes are dichotomous and are presented as alive or dead 10 years after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Josipa Glavas Tahtler, MD, Principal Investigator — Department of Anaesthesiology, Resuscitation and ICU, Osijek University Hospital,

IPD SHARING:
Plan to Share IPD: No
data may be shared upon request from researchers.

REFERENCES:
- [Background] Beguinot M, Monrigal E, Kwiatkowski F, Ginzac A, Joly D, Gayraud G, Le Bouedec G, Gimbergues P. Continuous Wound Infiltration With Ropivacaine After Mastectomy: A Randomized Controlled Trial. J Surg Res. 2020 Oct;254:318-326. doi: 10.1016/j.jss.2020.05.006. Epub 2020 Jun 5. PMID 32512380
- [Background] Kaur U, Shamshery C, Agarwal A, Prakash N, Valiveru RC, Mishra P. Evaluation of postoperative pain in patients undergoing modified radical mastectomy with pectoralis or serratus-intercostal fascial plane blocks. Korean J Anesthesiol. 2020 Oct;73(5):425-433. doi: 10.4097/kja.20159. Epub 2020 Sep 24. PMID 32987492
- [Background] Li R, Xiao C, Liu H, Huang Y, Dilger JP, Lin J. Effects of local anesthetics on breast cancer cell viability and migration. BMC Cancer. 2018 Jun 19;18(1):666. doi: 10.1186/s12885-018-4576-2. PMID 29914426
- [Background] Chen JL, Liu ST, Huang SM, Wu ZF. Apoptosis, Proliferation, and Autophagy Are Involved in Local Anesthetic-Induced Cytotoxicity of Human Breast Cancer Cells. Int J Mol Sci. 2022 Dec 7;23(24):15455. doi: 10.3390/ijms232415455. PMID 36555096
- [Background] Castelli V, Piroli A, Marinangeli F, d'Angelo M, Benedetti E, Ippoliti R, Zis P, Varrassi G, Giordano A, Paladini A, Cimini A. Local anesthetics counteract cell proliferation and migration of human triple-negative breast cancer and melanoma cells. J Cell Physiol. 2020 Apr;235(4):3474-3484. doi: 10.1002/jcp.29236. Epub 2019 Sep 20. PMID 31541469
- [Background] Kwakye AK, Kampo S, Lv J, Ramzan MN, Richard SA, Falagan AA, Agudogo J, Atito-Narh E, Yan Q, Wen QP. Levobupivacaine inhibits proliferation and promotes apoptosis of breast cancer cells by suppressing the PI3K/Akt/mTOR signalling pathway. BMC Res Notes. 2020 Aug 17;13(1):386. doi: 10.1186/s13104-020-05191-2. PMID 32807213
- [Background] Klein I, Kalichman L, Chen N, Susmallian S. Effect of physical activity levels on oncological breast surgery recovery: a prospective cohort study. Sci Rep. 2021 May 17;11(1):10432. doi: 10.1038/s41598-021-89908-8. PMID 34002007
- [Background] Meerkerk CDA, Chargi N, de Jong PA, van den Bos F, de Bree R. Sarcopenia measured with handgrip strength and skeletal muscle mass to assess frailty in older patients with head and neck cancer. J Geriatr Oncol. 2021 Apr;12(3):434-440. doi: 10.1016/j.jgo.2020.10.002. Epub 2020 Oct 13. PMID 33067163
- [Derived] Glavas Tahtler J, Djapic D, Neferanovic M, Miletic J, Milosevic M, Kralik K, Neskovic N, Tomas I, Mesaric D, Marjanovic K, Rajc J, Orkic Z, Cicvaric A, Kvolik S. Long-Term Outcomes of Breast Cancer Patients Receiving Levobupivacaine Wound Infiltration or Diclofenac for Postoperative Pain Relief. Pharmaceutics. 2023 Aug 23;15(9):2183. doi: 10.3390/pharmaceutics15092183. PMID 37765154